CLINICAL TRIAL: NCT05175313
Title: Transthoracic Ultrasonography Findings and Their Relation to Spirometric Indices in Patients With Obstructive and Restrictive Respiratory Diseases
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sohag University (Other)
Collaborators: Cairo University (Other)
Responsible Party: Principal Investigator, Esraa Faragallah Abdelaal, assistant lecturer, Sohag University
Other Study IDs: Soh-Med-21-12-15
Record Dates: First submitted 2021-12-14; First posted 2022-01-03 (Actual); Last update posted 2023-04-12 (Actual); Status verified 2023-04

CONDITIONS: Lung Ultrasound; Spirometry; Respiratory Diseases; Diaphragm Ultrasound
MeSH Terms: conditions — Respiratory Tract Diseases | interventions — Spirometry

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- normal people: people who don't complain of respiratory diseases will be examined by chest ultrasound and pulmonary function test.
  Interventions: Radiation: transthoracic ultrasonography; Device: spirometry
- obstructive respiratory diseases: the patients who are diagnosed with either COPD or asthma.
  Interventions: Radiation: transthoracic ultrasonography; Device: spirometry
- restrictive respiratory diseases: patient with either ILD
  Interventions: Radiation: transthoracic ultrasonography; Device: spirometry

INTERVENTIONS:
Radiation: transthoracic ultrasonography — 1. lung ultrasonography
  2. Diaphragm and respiratory muscle ultrasound
  3. inferior vena cava ultrasound
Device: spirometry — pulmonary function test : FVC, FEV1, FEV1/FVC will be measured.

SUMMARY:
Evaluation of respiratory function is considered a crucial component in the assessment of patients with a wide range of respiratory diseases. Spirometry is considered a common method of measuring pulmonary function. Recently, Transthoracic ultrasound yields important diagnostic information within minutes. Respiratory muscle ultrasound is used to evaluate the anatomy and function of the respiratory system.

ELIGIBILITY:
Inclusion Criteria:

1 -age >18 years 2-patients diagnosed with COPD or asthma. 3-patients diagnosed with ILD or any other restrictive lung diseases. 4-normal people.

Exclusion Criteria:

1. age <18 years old.
2. critically ill patients in intensive care units.
3. patients with neurological diseases.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: COPD: include patients with chronic bronchitis and emphysema. asthma: patients with paroxysmal attacks of chest tightness .wheezes and cough. ILD(interstitial lung diseases )
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-06 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
investigate the correlation between transthoracic ultrasonography findings and their relation to spirometric indices in patients with different respiratory diseases. | 6months
  we will study the degree of change in lung ultrasound, diaphragm, and respiratory muscles ultrasound, inferior vena cava ultrasound in obstructive and restrictive respiratory diseases .also, we find their correlation with spirometric indices in these diseases.

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag university hospital, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Santana PV, Cardenas LZ, Albuquerque ALP, Carvalho CRR, Caruso P. Diaphragmatic ultrasound: a review of its methodological aspects and clinical uses. J Bras Pneumol. 2020 Nov 20;46(6):e20200064. doi: 10.36416/1806-3756/e20200064. eCollection 2020. PMID 33237154
- [Background] Smargiassi A, Inchingolo R, Tagliaboschi L, Di Marco Berardino A, Valente S, Corbo GM. Ultrasonographic assessment of the diaphragm in chronic obstructive pulmonary disease patients: relationships with pulmonary function and the influence of body composition - a pilot study. Respiration. 2014;87(5):364-71. doi: 10.1159/000358564. Epub 2014 Apr 11. PMID 24732295
- [Background] O'Hara DN, Pavlov A, Taub E, Ahmad S. Ultrasonographic modeling of diaphragm function: A novel approach to respiratory assessment. PLoS One. 2020 Mar 12;15(3):e0229972. doi: 10.1371/journal.pone.0229972. eCollection 2020. PMID 32163474
- [Background] Santana PV, Cardenas LZ, de Albuquerque ALP, de Carvalho CRR, Caruso P. Diaphragmatic ultrasound findings correlate with dyspnea, exercise tolerance, health-related quality of life and lung function in patients with fibrotic interstitial lung disease. BMC Pulm Med. 2019 Oct 21;19(1):183. doi: 10.1186/s12890-019-0936-1. PMID 31638951
- [Background] Zanforlin A, Giannuzzi R, Nardini S, Testa A, Soldati G, Copetti R, Marchetti G, Valente S, Inchingolo R, Smargiassi A. The role of chest ultrasonography in the management of respiratory diseases: document I. Multidiscip Respir Med. 2013 Aug 9;8(1):54. doi: 10.1186/2049-6958-8-54. PMID 23937880